CLINICAL TRIAL: NCT05841875
Title: Efficacy and Safety of a Protocol Using C-reactive Protein to Guide Antibiotic Therapy Applied Through a Digital Clinical Decision Support Tool: a Randomized Clinical Trial
Brief Title: Efficacy and Safety of a Protocol Using C-reactive Protein to Guide Antibiotic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); FAPEMIG - FundaÃ§Ã£o de Amparo a Pesquisa do Estado de Minas Gerais (Unknown)
Responsible Party: Principal Investigator, Vandack Alencar Nobre, Clinical Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO.RAP
Record Dates: First submitted 2023-03-28; First posted 2023-05-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Systemic Infection
Keywords: Systemic infection; Sepsis; Biomarkers; C reactive protein; Antibiotic; Antibiotic stewardship
MeSH Terms: conditions — Toxemia; Sepsis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - C reactive protein (Experimental): For patients in the intervention group, attending physicians will be encouraged to follow an algorithm that uses clinical variables and serum CRP levels to guide the duration of antibiotic therapy. The peak CRP is defined as the highest value recorded within the first 72 hours of treatment.
  Antibiotic therapy discontinuation will be encouraged under the following conditions:
  If the peak CRP is below 100 mg/L: Consider stopping antibiotics when CRP falls below 35 mg/L, with a minimum treatment duration of 3 days.
  If the peak CRP is above 100 mg/L or the patient meets criteria for sepsis or septic shock: Consider stopping antibiotics when CRP has decreased by 50%, after a minimum of 5 days.
  If the patient does not meet the CRP criteria: Antibiotic discontinuation will be recommended after 5-7 days, provided there is clinical improvement.
  Interventions: Other: C reactive protein algorithm
- Control group: Best practice (No Intervention): For patients in the control group, the attending physician will be encouraged to determine the duration of antimicrobial therapy based on the best available evidence, taking into account the most likely infectious focus and the patient's clinical response. These recommendations will be guided by international society guidelines and established best practices for antibiotic therapy.
  Additionally, it is recommended that CRP monitoring in the control group be discontinued after 72 hours of antibiotic therapy, as this period is considered sufficient for using CRP as a biomarker to assist in diagnosing the infectious condition.

INTERVENTIONS:
Other: C reactive protein algorithm — Antibiotic therapy discontinuation will be encouraged under the following conditions:
  If the peak CRP is below 100 mg/L: Consider stopping antibiotics when CRP falls below 35 mg/L, with a minimum treatment duration of 3 days.
  If the peak CRP is above 100 mg/L or the patient meets criteria for sepsis or septic shock: Consider stopping antibiotics when CRP has decreased by 50%, after a minimum of 5 days.
  If the patient does not meet the CRP criteria: Antibiotic discontinuation will be recommended after 5-7 days, provided there is clinical improvement.
  Before discontinuing antibiotic therapy, physicians should confirm that the patient is clinically improving, with no signs of a persistent infectious focus. Additionally, they will be encouraged to verify that the Sequential Organ Failure Assessment (SOFA) score is stable or decreasing. These factors will assist in determining the appropriateness of stopping antibiotics.
  Arms: Intervention group - C reactive protein

SUMMARY:
The growing resistance of microorganisms to antimicrobials is a major threat to public health nowadays. Reducing the consumption of antibiotics is one of the main strategies to control this issue. Protocols using biomarkers to guide antimicrobial therapy have been studied, with promising results in safely reducing patient exposure to these drugs by reducing duration of treatments. Procalcitonin (PCT) and C-reactive protein (CRP) represent the most promising biomarkers in this context. Although less studied, CRP has the potential advantages of lower cost and wide availability when compared to PCT. However, decision algorithms involving biomarkers proposed in studies published so far are very far from daily medical practice in hospitals, mainly because there is poor accessibility to these protocols, and because most of them do not contemplate each patients clinical variables. The objective of this project is to evaluate the efficacy and safety of a multimodal protocol using clinical variables and the CRP value to guide antibiotic therapy in hospitalized patients. This protocol will be applied diretcly by the assistant medical teams through a digital clinical decision support tool available in the form of an application for mobile devices developed by the research team.

DETAILED DESCRIPTION:
The research team will perform a randomized, controlled, concurrent, open, single-center clinical trial. The proposed intervention is the application of a protocol that uses clinical variables and the CRP value to guide the duration of antibiotic therapy in patients with suspected or confirmed bacterial infection. As for the control group, the duration of antibiotic therapy will be suggested according to the best available evidence, considering the primary site of infection and other characteristics of this process. For both groups, the study protocol will be applied through a digital application for use on smartphones or tablets, developed specifically for this project. Participants will be adults admitted to the internal medicine ward of the Hospital das Clínicas of the Federal University of Minas Gerais (HC-UFMG), for whom the assistant physician team has started antibiotic therapy in the last 72 hours. Patients will be allocated after signing a free and informed consent form. Follow-up will be carried out until hospital discharge, death or 90 days, whichever occurs first. The project was submitted for consideration to the Research Ethics Committee of the Federal University of Minas Gerais (COEP-UFMG) and approved. As primary outcome, the duration of antibiotic therapy will be evaluated for the infectious episode that motivated inclusion in the study. Duration of antibiotic therapy will be measured by antimicrobial days (defined by the aggregate of days a specific antimicrobial agent was administered to an individual patient) per 1000 present days (defined by the length of time during which a given patient is at risk for antimicrobial exposure at a given institution). As secondary outcomes, the investigators will assess total exposure to antimicrobials, antibiotic-free days, user satisfaction after using the digital tool, protocol adherence rate, length of stay, estimated cost of antimicrobial therapy, all-cause hospital mortality, therapeutic failure, reinfection rate, subsequent infections with multidrug-resistant microorganisms, Clostridioides difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age,
* Clinical suspicion or microbiological confirmation of bacterial infection, with initiation of antibiotic therapy in the last 72 hours.
* Signing of the free and informed consent term by the patient or companion if the patient is unable to sign it (Annex 1).
* Patient admitted to the unit participating in the study.

Exclusion Criteria:

* HIV-infected patients with a CD4 count < 200 cells/mm3; neutropenic with neutrophil count < 500 cells/mm3; solid organ or bone marrow transplants; patients who received chemotherapy in the last 14 days at high risk of febrile neutropenia (> 20%), defined by the assistant team responsible for the treatment of the neoplasm; use of immunosuppressants, such as cyclophosphamide, azathioprine, cyclosporine, rituximab, tacrolimus, sirolimus or TNF inhibitors; use of corticosteroid therapy at a dose greater than 0.5mg/Kg of prednisone (or equivalent) over the last 30 days or pulse therapy in the last 14 days with these drugs; primary immunodeficiency (eg, X-linked agammaglobulinemia, common variable immunodeficiency) or patients with another condition that determines a clear impairment of immunological defenses, whether humoral, cellular or mixed.
* Conditions that require prolonged antibiotic therapy (infective endocarditis, necrotizing pneumonia, deep abscesses, osteomyelitis, complicated soft tissue infections, S. aureus bacteremia, among others), identified before randomization (ie, up to 72 hours of antibiotic therapy) .
* Patients with the perspective of hospital discharge in less than 72 hours from inclusion.
* Patients in exclusive palliative care.
* Patients with life expectancy < 24h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic therapy | From enrollment to the end of treatment.
  Duration of antibiotic therapy for the index infectious episode (the one that prompted inclusion in the study), measured in days.

SECONDARY OUTCOMES:
Total exposure to antimicrobials | 90 days
  Total antimicrobial exposure, defined as the number of days of antibiotic exposure considering all therapeutic cycles during patient follow-up, measured in Antimicrobial days / days of follow-up x 1,000. Antimicrobial days = total number of days antibiotics were given. If a patient is on 2 antibiotics, both are counted (i.e., the number of days for both drugs are added together). Days of follow-up = sum of days of follow-up in the study.
Antibiotic-free days | 90 days
  Defined by the ratio of the number of days of follow-up without the use of antibiotics by the number of days of follow-up in total, corrected by a denominator of 100.
Length of hospital stay | 90 days
  Measured in days.
Cost estimate of antimicrobial therapy. | 2 years
  Considering Brazilian market prices.
Adherence rate to the protocol in both the intervention and control groups. | 90 days
  The research team will closely monitor the daily progress of patients in each group, and will actively encourage adherence to the protocol associated with the respective group. For the intervention group, this may involve explaining the benefits of following the new algorithm, while for the control group, it may focus on adherence to the standard care. Any deviations from the algorithm will be noted for analysis.
All-cause 90 days mortality | 90 days
  All-cause 90 days mortality.
Therapeutic failure | 2 days
  Defined as persistence or recurrence of signs and symptoms of the same focus of infection that motivates resumption of antibiotic therapy in less than 48 hours after suspension.
Reinfection rate | 90 days
  Defined as a new episode of infection with a different focus or with isolation of new microorganisms or after 48 hours of discontinuation of antibiotic therapy directed at the initial infectious condition.
Subsequent infections by multidrug-resistant microorganisms | 90 days
  Measured by the ratio of cultured isolates per 100 patients.
Clostridioides difficile infection | 90 days
  Measured by diagnostic methods avaiable in Hospital das Clínicas da Universidade Federal de Minas Gerais.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The project will collect individual clinical and laboratory data from 200 patients, extracted from electronic medical records via the Aplicativo de Gestão para Hospitais Universitários (AGHU, 2009) and laboratory results from the MatrixNet system (MATRIXSAUDE, 2020). In addition, 3 to 5 serum aliquots of 0.5 ml each will be collected from each patient after informed consent is obtained. These aliquots will be stored for potential future analyses by the research team. Clinical and laboratory data will be securely stored using the Research Electronic Data Capture (REDCap) platform (Vanderbilt University, Nashville, USA, 2004). The serum samples will be preserved in a -80°C freezer in a biorepository that complies with the Institutional Biorepository Regulations. The biorepository will be housed at the School of Medicine, Federal University of Minas Gerais (UFMG), located at Av. Prof. Alfredo Balena, 190, Belo Horizonte - MG, CEP 30130-100.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Initially, the database generated by this project will remain restricted to the research team. Data sharing is anticipated at the time of associated publications, following proper anonymization of patient information. Data may be shared with journal editors or reviewers as part of the manuscript evaluation process, in compliance with journal requirements.
Access Criteria: Access to the scientific data will be limited to the research team via a permission-based system that requires login credentials. The serum samples stored in the biorepository will be similarly restricted, with access controlled in compliance with the Institutional Biorepository Regulations of the hosting institution. All data will be de-identified prior to sharing or distribution. A certificate of confidentiality will be included as part of the Informed Consent process to further safeguard participants privacy and rights.

REFERENCES:
- [Background] Borges I, Carneiro R, Bergo R, Martins L, Colosimo E, Oliveira C, Saturnino S, Andrade MV, Ravetti C, Nobre V; NIIMI - Nucleo Interdisciplinar de Investigacao em Medicina Intensiva. Duration of antibiotic therapy in critically ill patients: a randomized controlled trial of a clinical and C-reactive protein-based protocol versus an evidence-based best practice strategy without biomarkers. Crit Care. 2020 Jun 1;24(1):281. doi: 10.1186/s13054-020-02946-y. PMID 32487263
- [Derived] Rezende VMLR, Borges IN, Ravetti CG, De Souza RP, Vassalo PF, Caldas ACP, Gatto FR, Okamura GH, Lacerda RLB, Povoa PR, Nobre V. Efficacy and safety of an algorithm using C-reactive protein to guide antibiotic therapy applied through a digital clinical decision support system: a study protocol for a randomised controlled clinical trial. BMJ Open. 2025 Jan 27;15(1):e084981. doi: 10.1136/bmjopen-2024-084981. PMID 39870501